CLINICAL TRIAL: NCT04385147
Title: The Status of Advanced Endoscopy in the Era of COVID-19: a Multicenter Study
Brief Title: Advanced Endoscopy During COVID-19
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Collaborators: Helwan University (Other); National Liver Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mohamed Alboraie, Lecturer of medicine and gastroenterology, Al-Azhar University
Other Study IDs: Global-Endo-COVID
Record Dates: First submitted 2020-05-11; First posted 2020-05-12 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Cholangitis, Secondary Biliary; Cholangiocarcinoma; Obstructive Jaundice; Pancreas Cancer; COVID-19; SARS-CoV-2
Keywords: Obstructive Jaundice; Cholangitis; Pancreas Cancer; COVID-19; SARS-CoV-2; esophagogastroduodenoscopy; Endoscopy; Endoscopic retrograde cholangiopancreatography; Endoscopic ultrasound
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Cholangiocarcinoma; Jaundice, Obstructive; Pancreatic Neoplasms; COVID-19; Cholangitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERCP: Patients who will have endoscopic retrograde cholangiopancreatography
  Interventions: Other: Endoscopic management according to standard of care
- EUS: Patients who will have endoscopic ultrasound
  Interventions: Other: Endoscopic management according to standard of care

INTERVENTIONS:
Other: Endoscopic management according to standard of care — Endoscopic management according to standard of care by ERCP or EUS according to the indication in each case

SUMMARY:
In this study, investigators aim to explore the status of advanced endoscopy in different endoscopy units all over the world.

DETAILED DESCRIPTION:
In this study, investigators aim to explore the status of advanced endoscopy (endoscopic retrograde cholangiopancreatography and endoscopic ultrasound on a global level) in different endoscopy units all over the world, to report the characteristics of patients presented to these units and their procedure details.

evaluate the validity of different GI societies recommendations applied in different GI endoscopy units on the prevention of SARS-CoV-2 nosocomial transmission and the overall impact of this recommendations on the service provided by each GI unit.

Target audience:

- Physicians performing advanced gastrointestinal endoscopies in different countries.

Objectives:

* Primary objective:

  1- To explore the status of advanced endoscopy (endoscopic retrograde cholangiopancreatography and endoscopic ultrasound on a global level) in different endoscopy units all over the world, to report the characteristics of patients presented to these units and their procedure details.
* Secondary objectives:

  1. Effect of COVID-19 precautions on procedure time, procedure success, complications and patient outcomes
  2. Effect of COVID-19 on working time and staff number

Process:

A questionnaire containing advanced endoscopy procedure details in different countries will be distributed via emails. Responses will be collected in an online platform and data will be analyzed to reveal the effect of SARS-CoV-2 pandemic on different aspects of advanced endoscopy practice in the studied countries.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for ERCP or EUS during the study period

Exclusion Criteria:

* Patients refusing to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with digestive disorders referred for ERCP or EUS during the study period in the participating centers
Sampling Method: Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-05 (Actual)

PRIMARY OUTCOMES:
Age, gender, nationality | 3 months
  Investigators will report the baseline demographic data (age, gender, nationality) of all patients.
Indication for procedure, status of SARS-CoV-2 infection | 3 months
  Investigators will report the baseline data clinical data (indication for procedure, status of SARS-CoV-2 infection) of all patients.
Complete blood count and liver functions tests | 3 months
  Investigators will report the baseline laboratory data (complete blood count and liver functions tests) of all patients.
procedure related complications | 3 months
  Investigators will report the procedure related complications.

SECONDARY OUTCOMES:
Effect of COVID-19 precautions on procedure time | 3 months
  Investigators will report wether the precautions lead to increase timing of the procedure
Effect of COVID-19 precautions on staff number | 3 months
  Investigators will report wether the precautions affected staff number (increased or decreased)

CONTACTS AND LOCATIONS:
Locations (5):
- Kings County Hospital Center, Brooklyn, NY, USA, Albertson, New York, United States
- Al-Azhar Univerisity, Cairo, Egypt
- University Medicine Greifswald, Greifswald, Germany
- 2- Hospital Guillermo Kaelin De la Fuente - EsSalud, Lima, Peru
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Investigators may share data after first publication